CLINICAL TRIAL: NCT00759551
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Study of the Efficacy, Safety, and Tolerability of TAK-536 in Patients With Mild to Moderate Uncomplicated Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan in Subjects With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-03-TL-536-002; U1111-1113-8708 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Hypertension
Keywords: Blood Pressure; Drug Therapy; Systolic Pressure; Diastolic Pressure; Vascular Diseases
MeSH Terms: conditions — Hypertension; Vascular Diseases | interventions — azilsartan; olmesartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Azilsartan 2.5 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 5 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 10 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 20 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- Olmesartan 20 mg QD (Active Comparator)
  Interventions: Drug: Olmesartan

INTERVENTIONS:
Drug: Azilsartan — Azilsartan 2.5 mg, tablets, orally, once daily and olmesartan placebo-matching capsules and tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 2.5 mg QD
Drug: Azilsartan — Azilsartan 5.0 mg, tablets, orally, once daily and olmesartan placebo-matching capsules and tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 5 mg QD
Drug: Azilsartan — Azilsartan 10 mg, tablets, orally, once daily and olmesartan placebo-matching capsules and tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 10 mg QD
Drug: Azilsartan — Azilsartan 20 mg, tablets, orally, once daily and olmesartan placebo-matching capsules and tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 20 mg QD
Drug: Azilsartan — Azilsartan 40 mg, tablets, orally, once daily and olmesartan placebo-matching capsules and tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 40 mg QD
Drug: Placebo — Azilsartan placebo-matching tablets, orally, once daily and olmesartan placebo-matching capsules, orally, once daily for up to 8 weeks.
  Arms: Placebo QD
Drug: Olmesartan — Azilsartan placebo-matching tablets, orally, once daily and olmesartan 20 mg, capsules, orally, once daily for up to 8 weeks.
  Other Names: Benicar®; Olmetec®
  Arms: Olmesartan 20 mg QD

SUMMARY:
The purpose of this study is to determine the safety and efficacy of azilsartan, once daily (QD), in subjects with essential hypertension.

DETAILED DESCRIPTION:
According to the National Health and Nutrition Examination Survey, approximately 60 million people in the United States are hypertensive. Although no single risk factor is responsible for the development of hypertension, some of the many risk factors can be controlled, and some cannot. Controllable risk factors include weight gain, smoking, a sedentary lifestyle, poor eating habits, emotional stress, physical tension, sodium sensitivity, alcohol abuse, and use of oral contraceptives. Uncontrollable risk factors include family history, gender, age and race.

Hypertension is termed the "silent killer" because many patients are asymptomatic. Chronic hypertension causes extensive arterial wall damage, which allows cholesterol to adhere to the damaged endothelial lining and produces increased cardiac stress. Hypertension dramatically increases the risk of myocardial infarction, stroke, renal damage, impaired vision, heart failure and overall mortality. Angiotensin II receptor blockers are a class of drugs used for the treatment of hypertension that not only decrease blood pressure, but also likely contribute to protecting hypertensive individuals from cardiac events, strokes and loss of renal function.

Angiotensin II has significant physiological effects on tissues and organs throughout the body including vascular smooth muscle, adrenal cortex, kidney, and brain. Angiotensin II receptors are located on the plasma membrane of target cells to facilitate the rapid onset of angiotensin II. Three distinct subtypes of angiotensin II receptors have been identified: angiotensin II type-1 receptor, angiotensin type 2, and angiotensin type 4; and the relative proportion of each vary from tissue to tissue. The angiotensin II type-1 receptor subtype is expressed predominantly in vascular smooth muscle cells where activation by angiotensin II results in vasoconstriction, cell proliferation, fibrosis, and cellular hypertrophy. In contrast, angiotensin II type-2 receptor stimulation produces pharmacologic activities that are opposite to those that occur after angiotensin II type-1 receptor stimulation. The angiotensin II type-4 receptor has been reported to be expressed in the adrenals, brain, and myocardium, but its exact function remains unknown. It is not considered to play an important role in human pathogenesis.

TAK-536 (azilsartan) is a synthetic angiotensin II type-1 receptor antagonist being developed as a treatment for mild to moderate uncomplicated essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate uncomplicated essential hypertension (diastolic blood pressure between 95 and 114 mm Hg at Screening Day -7 and randomization visit).
* Female patients of childbearing potential must be nonpregnant and nonlactating, and utilizing an acceptable method of contraception.
* Has clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory unless the results are deemed not clinically significant for inclusion into this study by the investigator or sponsor.
* Is willing to discontinue current antihypertensive medications.

Exclusion Criteria:

* Has a decrease of more than or equal to 8 mm Hg in clinic diastolic blood pressure between Screening Day -7 and randomization visit.
* Is hypersensitive to angiotensin II receptor blockers.
* The patient has Grade 3 or 4 hypertensive retinopathy (Keith-Wagener scale).
* Has significant cardiac disease (eg, primary, hemodynamically significant cardiac valvular disease) other than mild to moderate uncomplicated hypertensive cardiovascular disease.
* Has taken, within 7 days prior to placebo run-in, or is expected to take, medications known to affect blood pressure, including the following:

  * Diuretics
  * Anti-hypertensives
  * Vasodilators
  * Tricyclic antidepressants
  * Monoamine oxidase inhibitors
  * Phenothiazines
  * Diet medications
  * Amphetamines or their derivatives
  * Thiazolidinediones
  * Lithium
  * Chronic use of common cold medications or nonsteroidal anti-inflammatory drugs including aspirin >325 mg/day or cyclooxygenase-2 inhibitors).
* Has a history of myocardial infarction complicated by heart failure, post-myocardial infarction angina, hypertensive encephalopathy, or cerebrovascular accident.
* Has clinically significant cardiac conduction defects (eg, 2nd or 3rd degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation or flutter).
* Has secondary hypertension of any etiology (eg, renal disease, pheochromocytoma, Cushing's syndrome).
* Has a history of collagen vascular disorder (eg systemic lupus erythematosus, scleroderma) within the last five years.
* Has an upper arm circumference less than 24 or greater than 42 cm.
* Works night (3rd) shift.
* Is non-compliant (less than 80%) with study medication during placebo run-in period.
* Has significant, moderate to severe renal dysfunction or disease (including renal artery stenosis).
* Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 2 years.
* Has a previous history of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study drug.
* Has Type I or Type II diabetes mellitus.
* Has an alanine transaminase or aspartate transaminase level of greater than 3 times the upper limit of normal, active liver disease, or jaundice.
* Is participating in another investigational study or has participated in an investigational study within 30 days prior to randomization.
* Has -any other serious disease or condition at Screening (or randomization) that would compromise patient safety, might affect life expectancy, or make it difficult to successfully manage and follow the patient according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2004-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in sitting clinic diastolic blood pressure. | Week 8 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in sitting clinic systolic blood pressure. | Weeks 2, 4, 6, and 8 or Final Visit
The change from Baseline in standing clinic diastolic blood pressure and systolic blood pressure. | Weeks 2, 4, 6, and 8 or Final Visit
Change from Baseline in diastolic blood pressure and systolic blood pressure as measured by ambulatory blood pressure monitoring. | Week 8 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda